CLINICAL TRIAL: NCT04901494
Title: Impact of SSRIs on the Rate of Progression of Patients With Mild Cognitive Impairment to Alzheimer's Disease Dementia and Other Neurodegenerative Dementias, With or Without Concurrent Use of Acetylcholinesterase Inhibitors
Brief Title: SSRI's and the Rate of Progression From MCI to Dementia
Status: Withdrawn | Type: Observational
Why Stopped: The PI is leaving the institution.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Maria Kataki, MD, PhD, Associate Professor of Clinical Neurology, Ohio State University
Other Study IDs: 2020H0375
Record Dates: First submitted 2021-05-11; First posted 2021-05-25 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment; Dementia; Alzheimer Disease
Keywords: SSRI
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SSRI for at least one year prior to the diagnosis of MCI: subjects with an initial diagnosis of MCI who were treated with an SSRI for at least one year prior to the diagnosis of MCI
  Interventions: Drug: SSRI
- SSRI at the time of diagnosis and treated with it for at least 6 months after the diagnosis of MCI: SSRI at the time of diagnosis and treated with it for at least 6 months after the diagnosis of MCI
  Interventions: Drug: SSRI
- Subjects without SSRI use: Subjects without SSRI use

INTERVENTIONS:
Drug: SSRI — Selective serotonin reuptake inhibitor
  Other Names: Selective serotonin reuptake inhibitor
  Groups: SSRI at the time of diagnosis and treated with it for at least 6 months after the diagnosis of MCI; SSRI for at least one year prior to the diagnosis of MCI

SUMMARY:
This trial is investigating if serotonin reuptake inhibitor (SSRI) use in Mild Cognitive Impairment (MCI) patients will lead to a lower rate of progression to dementia.

It's hypothesized that patients treated with an SSRI at the time of MCI diagnosis, without evidence of an active primary psychiatric condition other than neurocognitive disorder, will have a lower rate of progression to Alzheimer's disease dementia or to other types of dementia.

DETAILED DESCRIPTION:
Whether SSRIs affect the progression of MCI to dementia is not well studied with longitudinal prospectively collected date. Any decrease in the incidence of the progression of MCI to Alzheimer's dementia would be beneficial to patients.

This trial is investigating if serotonin reuptake inhibitor (SSRI) use in Mild Cognitive Impairment (MCI) patients will lead to a lower rate of progression to dementia.

This is a retrospective study of prospectively collected longitudinal data in patients followed at the Cognitive and Memory Disorders Center from 2010-2019. There are 3 arms: (1) subjects with an initial diagnosis of MCI who were treated with an SSRI for at least one year prior to the diagnosis of MCI (2) subjects with an initial diagnosis of MCI who were started on an SSRI at the time of diagnosis and treated with it for at least 6 months after the diagnosis of MCI and (3) subjects without SSRI use.

All the subjects have been evaluated based on a comprehensive standardized evaluation for the initial diagnosis and follow up over time. Chart reviews will be conducted on newly diagnosed MCI patients from 2010-2016 who have at least 2 years of annual follow up documented in their electronic medical record. Follow up visit notes through 2019 will be included in the review.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55+
2. Diagnosis of mild cognitive impairment.
3. One year treatment with an SSRI prior to diagnosis of MCI or six months treatment after diagnosis of MCI for the intervention groups. No treatment with an SSRI prior to the diagnosis of MCI or after the diagnosis of MCI for the control group.
4. A minimum of two annual follow up evaluations.

Exclusion Criteria:

1. Patients with CNS infection or inflammation
2. HIV
3. Syphilis
4. Patients with poorly controlled Epilepsy based on the opinion of the investigator.
5. Patients with space occupying lesions of the brain (glioma, meningioma, brain metastasis).
6. Patients with systemic inflammatory condition or cancer undergoing chemotherapy or on chronic immune modulatory treatments.
7. Blind patients that were not able to complete a cognitive assessment.
8. Patients with chronic pain who are on excluded pain medications.
9. Patients with Attention Deficit Disorder that require the use of stimulant medications.
10. Patients with Traumatic Brain Injury.
11. Patients with Cerebral Aneurysm Rupture.
12. Patients with chronic psychiatric conditions, unless in remission. Recurrent chronic psychiatric condition in relapse, chronic recurrent Major Depression in relapse, chronic recurrent bipolar disorder, chronic relapsing schizoaffective disorder and chronic recurrent anxiety disorder requiring chronic use of benzodiazepines are exclusionary.
13. Patients taking an excluded medication.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who meet the inclusion/exclusion criteria at the time of the initial diagnosis will be included in the review.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
SSRI rate of progression to dementia | 2010-2019
  1.To determine if subjects treated with an SSRI for at least one year prior to the diagnosis of MCI or at least 6 months after the diagnosis of MCI will (a) have a lower rate of progression to Alzheimer's disease dementia or (b) have a lower rate of progression to other dementia conditions (i.e. Lewy Body Dementia, Frontotemporal Dementia, Vascular Dementia, Normal Pressure Hydrocephalus, Parkinson Disease Dementia… etc) compared to subjects who are not treated with an SSRI.
SSRI and acetylcholinesterase inhibitor use progression to dementia | 2010-2019
  2.To determine if SSRI use in combination with acetylcholinesterase inhibitor use will affect the rate of progression to dementia.

SECONDARY OUTCOMES:
Rate of conversion from MCI to dementia and the other factors | 2010-2019
  1. To investigate correlations between the rate of conversion from MCI to dementia and other factors.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kataki, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No